CLINICAL TRIAL: NCT01297426
Title: Leptin Signaling in Humans
Brief Title: Leptin Signaling in Lean and Obese Humans
Acronym: Leptin signali
Status: Withdrawn | Type: Observational
Why Stopped: funding expired
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ENDA-013-10F
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Lean and obese, diabetic and non diabetics

SUMMARY:
Obesity does not respond to high circulating levels of the hormone leptin. This study is aiming at finding out why this happens and open new avenues for treatment of obesity.

DETAILED DESCRIPTION:
Ex vivo and in vitro identification and study of leptin signaling pathways in commercially available cell lines serum/ plasma samples and discarded tissues from humans.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* ages 18 to 65
* BMI ranges between 20 and 45 kg/m2

Exclusion Criteria:

* subjects requiring special diets
* history of illness other than obesity of diabetes
* taking medications known to influence glucose metabolism
* subjects with history of anaphylactic reaction or hypersensitivity to e. coli derived proteins or anesthetic agents
* women who are breastfeeding, pregnant or wanting to become pregnant
* subjects with bleeding dyscrasia or poor wound healing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetic or nondiabetic lean and obese subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Westerns / activation of signaling pathways (uo to two hours after treatment) | 04/01/2016

CONTACTS AND LOCATIONS:
Overall Officials: Christos Mantzoros, MD DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States